CLINICAL TRIAL: NCT06777732
Title: The Efficacy and Safety of Different Doses of Keverprazan Dual Therapy and Keverprazan-Based Bismuth Quadruple Therapy for Eradicating Helicobacter Pylori Infection: a Multicenter, Open, Randomized Controlled Study
Brief Title: The Efficacy and Safety of Keverprazan for Helicobacter Pylori Eradication
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20241217-09
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Amoxicillin; Furazolidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- standard dose keverprazan with high dose amoxicillin group (Active Comparator): Keverprazan Hydrochloride Tablets 20mg bid and Amoxicillin 1000mg tid for 14 days
  Interventions: Drug: Keverprazan; Drug: Amoxicillin
- low dose keverprazan with high dose amoxicillin group (Experimental): Keverprazan Hydrochloride Tablets 10mg bid and Amoxicillin 1000mg tid for 14 days
  Interventions: Drug: Keverprazan; Drug: Amoxicillin
- Keverprazan-based bismuth quadruple therapy (Experimental): Keverprazan Hydrochloride Tablets 20mg bid and Amoxicillin 1000mg bid and Furazolidone 100mg bid and Colloidal Bismuth Pectin 300mg bid for 14 days
  Interventions: Drug: Keverprazan; Drug: Amoxicillin; Drug: Furazolidone; Drug: Colloidal Bismuth Pectin

INTERVENTIONS:
Drug: Keverprazan — Potassium-competitive acid blocker
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: Furazolidone — Antibiotic for H. pylori eradication
  Arms: Keverprazan-based bismuth quadruple therapy
Drug: Colloidal Bismuth Pectin — Gastric mucosal protectant
  Arms: Keverprazan-based bismuth quadruple therapy

SUMMARY:
The purpose of this study was to compare the efficacy of 14-day eradication of Helicobacter pylori with different doses of Keverprazan combined with Amoxicillin dual therapy and Keverprazan-based bismuth quadruple therapy and compare the adverse reactions, compliance, and factors affecting the efficacy of eradication schemes among different groups.

DETAILED DESCRIPTION:
Helicobacter pylori infection is a major cause of gastrointestinal diseases, including peptic ulcers, chronic active gastritis, gastric mucosa-associated lymphoid tissue lymphoma, and fatal stomach cancer. At present, the infection rate of Helicobacter pylori in China is as high as 40.66%, and patients are often accompanied by a variety of upper digestive tract diseases, and about 1% of patients will develop malignant tumors. The Kyoto Global Consensus on Helicobacter Pylori Gastritis emphasizes that Hp gastritis is an infectious disease, HP-associated dyspepsia is an organic disease, and eradication of Hp can be used as a primary preventive measure for gastric cancer.At present, the first-line treatment for Hp eradication is a quadruple regimen of bismuth including proton pump inhibitor (PPI), bismuth agent and two antibacterial agents. However, its radical treatment of Hp still has limitations, mainly including increased side effects related to bismuth use and poor medication compliance. Clarithromycin and metronidazole have high drug resistance and high drug cost. Compared to H. pylori which is highly resistant to clarithromycin and metronidazole, resistance to amoxicillin and furazolidone in China and other countries in the Asia-Pacific region remains low.In recent years, the efficacy of high-dose amoxicillin regimen in eradicating H. pylori has been established, and its eradication rate and adverse reactions are similar to that of bismuth quadruple regimen, with better compliance and lower treatment cost. Potassium competitive acid blocker (P-CAB) is a new generation of acid suppressors. Compared with PPI, P-CAB has stronger acid inhibition effect, rapid onset, no acid activation, no influence of CYP2C19 genotype, long half-life, and better night acid inhibition than PPI.Meta-analyses have shown that P-CAB has a higher Helicobacter pylori eradication rate than PPI (90.2% vs. 75.5%). Keverprazan is a new type of potassium competitive acid blocker, whose acid inhibition is not affected by the environmental PH value, and has a more rapid and sustained acid inhibition effect. Keverprazan 20mg has a stable and lasting inhibitory effect on gastric acid. Several clinical studies have shown that Keverprazan is no less effective than lansoprazole in the treatment of reflux esophagitis and duodenal ulcer. The objective of this study was to evaluate the clinical efficacy of different doses of Keverprazan combined therapy and Keverprazan based bismuth quadruple therapy in the eradication of Helicobacter pylori infection. The three programs were compared from the aspects of eradication rate, compliance, adverse reactions and treatment cost, so as to provide reference and basis for the selection of Hp eradication programs, in order to further improve the effectiveness, safety and economy of Hp eradication and reduce the drug resistance of Hp.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65
2. Patients who tested positive for H. pylori by 13C or 14C breath test and have not received previous eradication therapy
3. Voluntarily join the trial and sign the informed consent form.

Exclusion Criteria:

1. Allergic to the study drug (e.g. penicillin allergy)
2. Recent bleeding or within 4 weeks of bleeding history in the stomach or duodenum
3. Patients who have previously received eradication therapy for Helicobacter pylori
4. Use antibiotics or bismuth medication 4 weeks before starting the study；use P-CAB or PPI 2 weeks before starting the study
5. Patients who have had surgery on the stomach or intestines, which affects the drug's metabolism
6. Pregnant or lactating women
7. Patients with other serious physiological or psychological conditions, or those with liver or kidney dysfunction
8. Patients with Zollinger-Ellison syndrome, gastric mucosal-associated lymphoid tissue lymphoma (MALT), or malignant tumors
9. Patients with glucose-6-phosphate dehydrogenase (G-6PD) deficiency, peptic ulcer disease, or bronchial asthma
10. Patients with concomitant medications including azatanavir or lopinavir, tricyclic antidepressants, levodopa, paracetamol, codeine phosphate/dextromethorphan, monoamine oxidase inhibitors, tramadol, etc.
11. Other factors that the investigator considers unsuitable for participation in the study, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Within 7 days after completion of therapy
  Adverse drug reactions are classified into six types: dose-related, non-dose-related, dose-related and time-related, time-related, withdrawal, and failure of therapy.

SECONDARY OUTCOMES:
Helicobacter pylori eradication rate | four to six weeks after completion of the medication
  Helicobacter pylori Eradication will be determined by ¹³C-urea breath test four to six weeks after completion of the medication. The eradication rates will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.

IPD SHARING:
Plan to Share IPD: No